CLINICAL TRIAL: NCT04423900
Title: Smart Phone-Based Application for Evaluation and Rehabilitation of HindFoot Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: YeditepeFTR
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Achilles Tendinopathy; Plantar Fascitis; Feet Pes Cavus; Feet Pes Planus (Flatfoot); Foot Diseases
Keywords: telerehabilitation; hind foot pain; plantar fasciitis; achilles tendinopathy; smart phone
MeSH Terms: conditions — Talipes Cavus; Clubfoot; Foot Diseases; Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: One hundred twenty patients aged 18-75 years, diagnosed as Plantar fasciitis and Achilles Tendinopathy by an Orthopedic surgeon, will be included. Patients will be randomly divided into three groups according to inclusion criteria.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Plantar Fasciitis App Exercise Group (Experimental): Video simulation of patient education (definition of the disease, risk factors, lifestyle modifications, prevention methods) will be performed to people via smart phone app application. Individuals will receive feedback after completing the training program and will then be included in the exercise program. The mobile application provides feedback so that the exercise program (stretching, strengthening, self-myofascial relaxation exercises) determined according to the diagnosis of the patients is performed by the patients at twice a day for eight weeks.
  Interventions: Diagnostic Test: smart phone application
- Achilles Tendinopathy App Exercise Group (Experimental): Video simulation of patient education (definition of the disease, risk factors, lifestyle modifications, prevention methods) will be performed to people via smart phone app application. Individuals will receive feedback after completing the training program and will then be included in the exercise program. The mobile application provides feedback so that the exercise program (stretching, strengthening, self-myofascial relaxation exercises) determined according to the diagnosis of the patients is performed by the patients at twice a day for eight weeks.
  Interventions: Diagnostic Test: smart phone application
- Plantar Fasciitis Home Exercise Group (Experimental): Patients will learn the exercises by the physiotherapist in the clinic. Patients will be included in the training program (stretching, strengthening, self-myofascial release exercises) -only once. Then, patients will do this program at their home twice a day for eight weeks.
  Interventions: Diagnostic Test: smart phone application
- Achilles Tendinopathy Home Exercise Group (Experimental): Patients will learn the exercises by the physiotherapist in the clinic. Patients will be included in the training program (stretching, strengthening, self-myofascial release exercises) -only once. Then, patients will do this program at their home twice a day for eight weeks.
  Interventions: Diagnostic Test: smart phone application
- Plantar Fasciitis Conventional Physiotherapy Group (Experimental): In this group, patients will first be included in the patient education and exercises program in the clinic-only once. Mulligan Concept - Manual Therapy and Compressive myofascial relaxation methods will be applied to the individuals who have completed the patient training program by the physiotherapist. Patients will participate in the rehabilitation program twice a week for eight weeks. These patients will perform their home exercises twice daily and for eight weeks.
  Interventions: Diagnostic Test: smart phone application
- Achilles Tendinopathy Conventional Physiotherapy Group (Experimental): In this group, patients will first be included in the patient education and exercises program in the clinic-only once. Mulligan Concept - Manual Therapy and Compressive myofascial relaxation methods will be applied to the individuals who have completed the patient training program by the physiotherapist. Patients will participate in the rehabilitation program twice a week for eight weeks. These patients will perform their home exercises twice daily and for eight weeks.
  Interventions: Diagnostic Test: smart phone application

INTERVENTIONS:
Diagnostic Test: smart phone application — Participants will be asked to provide information about their sociodemographic characteristics, chronic diseases, the history of the ankle injury, trauma, and surgery, the severity of the foot pain via using the mobile application.The app will be downloaded from the Google Play Store and available offline. Information from the patient will be stored in an SQLite database.The usability test will be carried out on the mobile application so that the latest releases contain clear, effective, loyal to the strategy, and easily understood messages by the intended audience and do not produce unwanted responses.Direct observation, individual interviews, and satisfaction surveys will be used to identify areas of improvement in a cross-sectional manner.Investigation of pes cavus, pes planus and ankle range of motion will be determined by image processing.All data can be analyzed and stored by Heel Analysis Systems established on an external server.The data will be transferred securely over HTTPS.

SUMMARY:
This randomized controlled study aims to evaluate the status of the individuals with hindfoot pain and to recommend preventive precautions and appropriate exercise programs with Smart Phone-Based Applications. Additionally, to compare the results of patients who attended through mobile applications (Achilles Tendinopathy and Plantar Fasciitis) with the results of patients included in the hands-on program.

DETAILED DESCRIPTION:
Foot pain is common in the general population, with prevalence estimates ranging from 17 to 30% . A systematic review concluded that nearly one-quarter of adults over age 45 experience frequent foot pain. Foot pain has been associated with poor balance, gait problems, the limitation of daily living activities, and health-related quality of life. It has been reported that at least two-thirds of individuals experience moderate functional daily life problems .The etiology of hindfoot pain is mostly associated with Achilles Tendinopathy and Plantar Fasciitis, which are prevalent, affecting millions of people each year . Most cases of hindfoot pain if not treated, they will get worse with time and resistant symptoms. This is why to get more information on prevalence and risk factors in the general population is necessary to organize health care planning and the extent of clinical need.An increase in the use of digital technology and smart phones globally with mobile applications provide an alternative solution to the planning of primary health care services. In the US, approximately 90% of adults have a mobile phone, and 58% of these prefer smart phones, while in Turkey, 98% of adults use mobile phones, and 77% of them are smart phones owners. The popularity of smart phones provides opportunities for reaching information and giving skills to users through applications. These applications offer new opportunities for collecting, evaluating, and monitoring health information and have portability, the flexibility of use, and a width of the access area.With the concept of this approaching (using digital technologies,) several systematic reviews have examined digital programs using for different health conditions/ pathologies (paralysis, lack of balance/stabilization, cardiac disorders, and joint / extremity). A great deal of physiotherapy interventions for hindfoot pain includes electrotherapy agents, 'hands-on' therapy, stretching, and strengthening exercises. The exercise programs are an essential part of rehabilitation programs for hindfoot pain, and patients who involved in this exercise program also need to get feedback by physiotherapist. For this reason, the digital technology-based applications are considered to be contributive for follow-up exercise regularly and detecting the changes and progression. Additionally, to the best of our knowledge, a smartphone application research involving hindfoot pathology with suggesting assessment methods and including exercise program is not available in the literature. Thereby, the study aims to evaluate the status of the individuals with hindfoot pain and to recommend preventive precautions and appropriate exercise programs with Smart Phone-Based Applications and to compare the results of patients who attended through mobile applications (Achilles Tendinopathy and Plantar Fasciitis) with the results of patients included in the hands-on program.

ELIGIBILITY:
Inclusion Criteria:

* Pain in the heel and surrounding area
* Have given consent to be a volunteer for participating to the study
* 18 years and older
* Ability to use a smartphone

Exclusion Criteria:

* Having foot and ankle injury and surgery in the last three months
* Have received physiotherapy or local injection before randomization
* Having major pathologies during the rehabilitation program (severe heart and neuropsychiatric disorders, complicated diabetes mellitus)
* Neoplastic formation in the foot-ankle region
* Vision problem
* Night pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Feiss Line test | 8 weeks
  Feiss Line is an ankle examination procedure that tests for pes planus, flatfoot, fallen medial longitundinal arch.Patient should be standing with weight distributed evenly.
  The examiner uses a marker to mark the inferior apex of medial malleolus and medial surface of the base of the base of the 1st metatarsal.
  The examiner draws a line connecting the two points. The examiner locates the the navicular tuberosity and marks it.
the Range of Motion of the ankle | 8 weeks
  Physiotherapist will measure the Range of Motion of the ankle by using Goniometer
Visual Analog Scale - Pain Assesment | 8 weeks
  Visual Analogue Scale (VAS) was used to estimate the severity of participants' first step (morning time) and activity pain. It consists of a line, usually 100 mm long, whose ends are labeled as the extremes (no pain and worst pain imaginable); the rest of the line is blank.

SECONDARY OUTCOMES:
Tampa Scale for Kinesiophobia | 8 weeks
  Tampa consists of 17 questions and is used in diseases associated with acute and chronic low back pain, fibromyalgia, and musculoskeletal injuries. The scale uses a 4-point Likert score (1 = Strongly disagree, 4 = Strongly agree). A total score is calculated after the reversal of items 4, 8, 12, and 16. The patients can have a total score of between 17-68. The higher the score indicates, the higher the kinesiophobia

OTHER OUTCOMES:
The Victorian Institute of Sport Assessment-Achilles Questionnaire | 8 weeks
  The VISA-A aims to evaluate the clinical severity of patients with chronic Achilles tendinopathy. It can be used to determine the patient's clinical severity and provide a guideline for treatments as well as for monitoring the effect of treatment. Robinson et al. designed the Victorian Institute of Sports Assessment-Achilles (VISA-A) questionnaire, as a region-specific functional questionnaire, to assess the severity of AT.6 It contains eight questions that cover the three domains of pain (questions 1-3), function (questions 5-7) and activity (questions 7 and 8). Scores are summed to give a total out of 100. An asymptomatic person would score 100. It has proven to be a valid and reliable instrument to measure disability in cross-cultural studies conducted in Turkey
Foot Function Index | 8 weeks
  FFI assessed pain, activity restriction, and disability. The pain subscale, which includes nine items, measures foot pain related to a variety of conditions. Various functional activities depending on foot problems were determined by the disability subscale, which also includes nine items. Activity restrictions due to foot problems were assessed with an activity limitation subscale containing five items. Higher scores indicate more pain, disability, and limited activity. In our study, the patients were asked to mark each category with a score between 0 and 10 about their pain, activity restriction, and disability level. All the categorized scores were collected, and a total score was noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Elif Tuğçe Çil, Istanbul, Europe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided